CLINICAL TRIAL: NCT03891472
Title: Clinical Phase II Clinical Study Evaluating the Toxicity and Efficacy of mFOLFIRINOX Associated With SBRT (Stereotactic Radiotherapy) in Patients With Unresectable Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Katarzyna Kuśnierz, Investigator, Medical University of Silesia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNW/0022/KB1/71/I/16
Record Dates: First submitted 2019-03-11; First posted 2019-03-27 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Cancer of Pancreas; Unresectable Pancreatic Cancer; Chemotherapy Effect; SBRT
Keywords: mFOLFIRINOX; SBRT; Unresectable Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Fluorouracil; Radiosurgery; Surgical Procedures, Operative; Pancreatectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Patients will receive initial chemotherapy, followed by evaluation of the response to the treatment, followed by SBRT, followed by chemotherapy.

INTERVENTIONS:
Drug: Patients will receive initial chemotherapy, followed by evaluation of the response to the treatment, followed by SBRT, followed by chemotherapy. — mFOLFIRINOX > SBRT > mFOLFIRINOX > Surgical Intervention
  Other Names: mFOLFIRINOX (Oxaliplatin, Irinotecan, Fluorouracil); SBRT (Stereotactic Body Radiation Therapy); Surgical Intervention (Pancreatectomy)

SUMMARY:
Primary goal:

Improvement of the therapeutic index by reducing the toxicity of treatment and increasing local control of the cancer process while evaluating the possibility of conversion to the surgical status.

Secondary targets:

* Survival rate (OS) assessment in patients treated with mFOLFIRINOX + SBRT
* Assessment of quality of life using questionnaires: EQ-5D, EORTC (QLQ-C30) and pancreatic cancer-specific QLQ PAS module 26
* Early toxicity <3 months after completion of SBRT treatment.
* Percentage of local control (1-year)

DETAILED DESCRIPTION:
STUDY PLAN Patients will receive initial mFOLFIRINOX (6 cycles) chemotherapy, followed by evaluation of the response to the treatment (imaging and laboratory testing) followed by SBRT, followed by mFOLFIRINOX chemotherapy.

In case of exclusion of disease progression after 10 weeks +/- 2 weeks after completion of SBRT, patients will be qualified to surgical treatment to attempt a radical surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signing informed consent for treatment.
2. Age> = 18 years.
3. Patients with histopathological diagnosis of adenocarcinoma of the pancreas.
4. Advanced disease referred to as locally advanced definitive non-resetable, non-metastatic pancreatic cancer.
5. No prior systemic treatment due to pancreatic adenocarcinoma
6. No prior radiotherapy in the abdominal area
7. No prior radical surgical treatment due to pancreatic adenocarcinoma (palliative surgical procedures such as bypass surgery or biliary tract surgery are acceptable).
8. ECOG 0 or 1.
9. Expected survival time in excess of 12 weeks.
10. Adequate organ performance based on laboratory blood tests.

Exclusion Criteria:

1. Patients diagnosed with other types of pancreatic cancer than adenocarcinomas (eg neuroendocrine cancer).
2. Advanced disease that allows primary surgical treatment.
3. Borderline pancreatic cancer (BRPC) disease.
4. The presence of metastases.
5. Previous systemic treatment because of pancreatic adenocarcinoma.
6. Preoperative radiotherapy in the abdominal area.
7. Previous radical surgery for pancreatic adenocarcinoma.
8. Large surgical procedure with the exception of diagnostic biopsies within the last 4 weeks after the start of treatment and / or patients who have not fully recovered after surgery.
9. Heart failure (NYHA Class II, III or IV)
10. Hemodynamic instability in the course of coronary and / or valvular heart disease and / or hypertension and / or other clinical conditions (eg uncontrolled diabetes mellitus).
11. Clinically relevant cardiac arrhythmias requiring treatment.
12. Stroke and / or myocardial infarction history within 6 months of inclusion.
13. Respiratory failure associated with other co-morbidities.
14. Serious psychiatric illnesses, which, in the researcher's opinion, could have a significant negative impact on the safety of the treatment.
15. Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.
16. Transplanted organ transplant including allogeneic bone marrow transplant.
17. Positive diagnosis for HBV or HCV indicating acute or chronic infection (for screening).
18. HIV infection.
19. The period of pregnancy and breastfeeding.
20. Alcoholism or drug abuse.
21. Limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Improvement of the therapeutic index. | 24 months.
  Improvement of the therapeutic index by reducing the toxicity of treatment and increasing local control of the cancer process while evaluating the possibility of conversion to the surgical status.
Improvement of the overall survival. | 60 months.
  Improvement of the overall survival by new treatment method.

CONTACTS AND LOCATIONS:
Locations (1):
- UCK Katowice, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided